CLINICAL TRIAL: NCT06344078
Title: Surgical Italian Guide for the Management of Complicated Acute Diverticulitis in Emergency Setting (SIGMA-D). A Prospective Observational Multicenter Study on Behalf of the Italian Society of Colorectal Surgery (SICCR).
Brief Title: Surgical Italian Guide for the Management of Complicated Acute Diverticulitis Emergency Setting (SIGMA-D). A Prospective Observational Multicenter Study on Behalf of the Italian Society of Colorectal Surgery (SICCR).
Acronym: SIGMA-D
Status: Recruiting | Type: Observational
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Principal Investigator, Donato F Altomare, DR FERRARA FRANCESCO, Societa Italiana di Chirurgia ColoRettale
Other Study IDs: SIGMA-d
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Acute Diverticulitis; Stoma Colostomy; Stoma Ileostomy
MeSH Terms: interventions — Anastomosis, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients operated for acute diverticulitis: patient with acute diverticulitis which are operated in urgency setting
  Interventions: Procedure: sigmoid resection and anastomosis / stoma

INTERVENTIONS:
Procedure: sigmoid resection and anastomosis / stoma — intestinal resection and recostruction or creation of stoma

SUMMARY:
This study will include data collected from surgical units performing emergency surgery in Italy during 2024, with a one-year follow-up period for each patient. Data for each center will be prospectively collected through a database filled out by the Italian Society of Colorectal Surgery (SICCR) members who participate to the study. Specific data will include: WSES diverticulitis classification, procedure timing, laparoscopic/converted procedures, rate of performed protection ileostomies or colostomies, rate and timing of Hartmann reversal or stoma closure, procedures with more than two operators, procedures with expert first operator, night or weekend procedures, and patients aged over 80. Postoperative data will focus on complication rates and mortality at one, six, and twelve months.

ELIGIBILITY:
Inclusion Criteria:

* 18 yo or older
* CT scan and WSES classification
* surgical intervention within 48 hours for acute diverticulitis

Exclusion Criteria:

* underaged
* conservative treatment for acute diverticulitis
* other treatment
* diagnosis of colorectal cancer at histology

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general population
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
adhesion to guidelines | 1 year follow-up
  assess whether Italian colorectal surgeons adhere to current guidelines, providing insights into the management of this disease.

SECONDARY OUTCOMES:
stoma reversal | 1 year follow-up
  understanding of the management of patients with stomas resulting from Hartmann's procedures or resection with primary anastomosis and protective stomas.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera universitaria paolo giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Undecided